CLINICAL TRIAL: NCT05169749
Title: The Effect of Preoperative Nursing Visit on Anxiety and Pain Level of Patients After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Yasemin Uslu, Asisst. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK 2018-16/33
Record Dates: First submitted 2021-11-29; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Nurse-Patient Relations
Keywords: Operating room nurse; Nursing visit; Laparoscopic surgery; Patient education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control-Service Nurse Group (Other): Patient education lasting 20-30 minutes was provided by the nurse who gives care in the surgical inpatient floor before the surgery. The nurse provided the patient's admission to the postoperative surgical inpatient floor and follow-up.
  Interventions: Procedure: Control-Service Nurse Group
- Experimental-Nursing Visiting Group (Experimental): The nursing visit was done by the operating room nurse who will be involved in the patient's surgery, and the patient education lasted 20-30 minutes. The nurse, who carried out the nursing visit, welcomed the patient in the operating room, was next to the patient before anesthesia, and followed the patient to the recovery room after surgery.
  Interventions: Procedure: Nursing Visiting Group

INTERVENTIONS:
Procedure: Control-Service Nurse Group — Processing Steps
  * The State-Trait Anxiety Inventory was applied before the patient education
  * The State Anxiety Inventory was applied after the education.
  * The pain was monitored in accordance with the surgical patient follow-up protocol for 24 hours postoperatively
  * The State Anxiety Inventory was applied again 24 hours after surgery.
  Arms: Control-Service Nurse Group
Procedure: Nursing Visiting Group — Processing Steps
  * The State-Trait Anxiety Inventory was applied before the patient education
  * The State Anxiety Inventory was applied after the education.
  * The pain was monitored in accordance with the surgical patient follow-up protocol for 24 hours postoperatively
  * The State Anxiety Inventory was applied again 24 hours after surgery.
  Arms: Experimental-Nursing Visiting Group

SUMMARY:
A nursing visit is a method used for psychological preparation and information of patients. During nursing visits, the operating room nurse visits the patient before the surgery, informs the patient about the surgical process and nursing care practices and gives education. The study was conducted to determine the effect of nursing visit before laparoscopic surgery on the anxiety and pain level of the patient in the postoperative period.

DETAILED DESCRIPTION:
In this study, a structured education program was created, the visiting nurse was ensured to be the nurse who is involved in the patient's surgery, and the levels of anxiety and pain were evaluated according to objective criteria in the postoperative period on the patient group planned for laparoscopic surgery.

The study was conducted with 135 patients, 72 in the experimental group and 63 in the control group. The website https://www.randomlists.com/random-letters was used during the randomization of the patients. The patients were randomly assigned to the experimental and control groups according to their sequence numbers.

For the standardization of patient education, an education booklet was prepared in line with the literature, and the final version was prepared by consulting experts. The experimental group was educated by visits of the operating room nurse. The control group was educated by the service nurse. Data were collected with state-trait anxiety inventory and visual analog scale.

Visual analog scale (VAS)- The scale, which is used to evaluate the pain intensity, aims to explain the patient's pain in numbers. The scale requires the patient to score the pain as the absence of pain starting from 0 (zero) and unbearable pain to be evaluated over 10 (ten) points Spielberger State-Trait Anxiety Inventory - Anxiety inventory was developed by Spielberg et al. in 1970 and adapted into Turkish by Oner and Le Compte in 1977. This inventory is a four-degree Likert type scale ranging from "Almost never" to "Almost always". In the state anxiety scale, the individual evaluates how he/she feels "right now". The total score obtained from each scale varies between 20 and 80. A high score indicates a high anxiety level, a low score indicates a low anxiety level The State-Trait Anxiety Inventory was applied before the patient education and the State Anxiety Inventory after the education. The pain was monitored in accordance with the surgical patient follow-up protocol for 24 hours postoperatively, and the State Anxiety Inventory was applied again 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were 18 years old and above
* who could speak Turkish and who were able to communicate
* underwent laparoscopic general surgery (such as laparoscopic cholecystectomy, colon, inguinal hernia, appendectomy, incisional hernia, sleeve gastrectomy) were included in the study.

Exclusion Criteria:

* Emergency and unplanned cases,
* patients transferred to the intensive care unit after surgery,
* patients with neurological or psychological problems were excluded from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in State Anxiety Level | Baseline to 24 hours postoperative
  State Anxiety Level is evaluated by Spielberger State-Trait Anxiety Inventory - This inventory is a four-degree Likert type scale ranging from "Almost never" to "Almost always". In the state anxiety scale, the individual evaluates how he/she feels "right now". The total score obtained from each scale varies between 20 and 80. A high score indicates a high anxiety level, a low score indicates a low anxiety level. Before, the patient education (before surgery) After, the education (before surgery) 24 hours after surgery.
Change in Pain Score | Baseline to 24 hours postoperative
  Pain score is evaluated by Visual analog scale (VAS). The scale, which is used to evaluate the pain intensity, aims to explain the patient's pain in numbers. The scale requires the patient to score the pain as the absence of pain starting from 0 (zero) and unbearable pain to be evaluated over 10 (ten) points. Immediately after surger: Every 1 hour and 15 minutes after being admitted to the surgical inpatient floor (15 minutes-30 minutes-45 minutes-60 minutes), every next 2 hours and 30 minutes (90 mins-120 mins-150 mins-180 mins), every next 4 hours (4th-5th-6th-7th hour), every next 4 hours (11th-15th-19th-24th hours). Data were collected between the zero and 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Uslu, Asisst Prof, Principal Investigator — Acıbadem Mehmet Ali Aydınlar Üniversitesi
Locations (1):
- Yasemin Uslu, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carter L, Evans T. Preoperative visiting: a role for theatre nurses. Br J Nurs. 1996 Feb 22-Mar 13;5(4):204, 206-7. doi: 10.12968/bjon.1996.5.4.204. PMID 8704447
- [Result] Coll AM, Ameen JR, Mead D. Postoperative pain assessment tools in day surgery: literature review. J Adv Nurs. 2004 Apr;46(2):124-33. doi: 10.1111/j.1365-2648.2003.02972.x. PMID 15056325
- [Result] Guo P, East L, Arthur A. A preoperative education intervention to reduce anxiety and improve recovery among Chinese cardiac patients: a randomized controlled trial. Int J Nurs Stud. 2012 Feb;49(2):129-37. doi: 10.1016/j.ijnurstu.2011.08.008. Epub 2011 Sep 22. PMID 21943828
- [Result] Marcus C. Strategies for improving the quality of verbal patient and family education: a review of the literature and creation of the EDUCATE model. Health Psychol Behav Med. 2014 Jan 1;2(1):482-495. doi: 10.1080/21642850.2014.900450. Epub 2014 Apr 28. PMID 25750796
- [Result] Sadati L, Pazouki A, Mehdizadeh A, Shoar S, Tamannaie Z, Chaichian S. Effect of preoperative nursing visit on preoperative anxiety and postoperative complications in candidates for laparoscopic cholecystectomy: a randomized clinical trial. Scand J Caring Sci. 2013 Dec;27(4):994-8. doi: 10.1111/scs.12022. Epub 2013 Jan 28. PMID 23350886
- [Derived] Aydal P, Uslu Y, Ulus B. The Effect of Preoperative Nursing Visit on Anxiety and Pain Level of Patients After Surgery. J Perianesth Nurs. 2023 Feb;38(1):96-101. doi: 10.1016/j.jopan.2022.05.086. Epub 2022 Aug 13. PMID 35970660